CLINICAL TRIAL: NCT00900848
Title: Traumatic Disruption of Iliofemoral Arterial Segment is Often Associated With Multiple Injuries, Massive Hemorrhage, State of Shock, and Loss of Blood Supply to the Ipsilateral Lower Extremity, as Well as With High Mortality
Brief Title: Posterior Tibial Artery Bypass for Iliofemoral Artery Injury Associated With Massive Blood Loss and Shock
Status: Completed | Type: Observational
Sponsor: The Second Hospital of Qinhuangdao (Other)
Responsible Party: Microsurgery, the Second hospital of Qinhuangdao
Other Study IDs: SHQ-0905-A
Record Dates: First submitted 2009-05-09; First posted 2009-05-13 (Estimated); Last update posted 2009-05-13 (Estimated); Status verified 2009-05

CONDITIONS: Iliofemoral Artery Injury; Shock
Keywords: Posterior tibial artery bypass; Iliofemoral artery injury; Shock; Reconstruction
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 8: 8 patients

SUMMARY:
Traumatic disruption of iliofemoral arterial segment is often associated with multiple injuries, massive hemorrhage, state of shock, and loss of blood supply to the ipsilateral lower extremity, as well as with high mortality.

The investigators describe a bypass technique. It can provide adequate blood supply to the lower extremity of the injury side. Due to a minimum amount of additional blood loss, it is a low risk procedure for salvage of the extremity and even patient's life.

DETAILED DESCRIPTION:
Patients were selected on the basis of the following: (1) closed injuries to the lower abdomen and/or pelvis; (2) serious hemorrhagic shock; (3) loss of blood supply to the ipsilateral lower extremity; (4) high-risk emergency artery reconstruction.

The instruments used to measure sensibility of the foot were the Semmes-Weinstein (SW) monofilament test 24 and the static two-point discrimination (2PD) test 25. The weight-bearing area of the first metatarsal head and the dorsum of the first metatarsal head were assessed. Active range of motion (ROM) of the hip, knee, and ankle joints was measured with a goniometer. The muscle strength was test using Medical Research Council (MRC) Scale. The cold intolerance of the leg was measured using the self-administered Cold Intolerance Severity Score (CISS) questionnaire 26. The maximum score is 100 and is grouped into 4 ranges (0-25, 26-50, 51-75, and 76-100) corresponding to mild, moderate, severe, and extreme severity, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. closed injuries to the lower abdomen and/or pelvis;
2. serious hemorrhagic shock;
3. loss of blood supply to the ipsilateral lower extremity;
4. high-risk emergency artery reconstruction.

Exclusion Criteria:

1. bleeding can be easily control through an open wound;
2. mild shock without life threatening conditions;
3. good blood supply to the ipsilateral lower extremity;
4. low-risk emergency artery reconstruction.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 8 patients
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2009-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xu Zhang, MD, Study Chair — The Second Hospital of Qinhuangdao